CLINICAL TRIAL: NCT01328899
Title: Feasibility Study of the PneumRx, Inc. Lung Volume Reduction Coil for the Treatment of Emphysema
Brief Title: Feasibility Study of PneumRx's Lung Volume Reduction Coil (LVRC)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Collaborators: PneumRx, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLN0011
Record Dates: First submitted 2011-04-01; First posted 2011-04-05 (Estimated); Last update posted 2021-07-21 (Actual); Status verified 2021-07

CONDITIONS: Emphysema
Keywords: Emphysema; COPD; RePneu
MeSH Terms: conditions — Emphysema; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Lung Volume Reduction Coil (LVRC) (Experimental): Lung Volume Reduction Coil (LVRC)
  Interventions: Device: Lung Volume Reduction Coil (LVRC) (PneumRx's)

INTERVENTIONS:
Device: Lung Volume Reduction Coil (LVRC) (PneumRx's) — Lung Volume Reduction Coil
  Other Names: Lung Volume Reduction Device (LVRD)

SUMMARY:
This is a multicenter single arm open label study. The primary objective is to evaluate the safety and effectiveness of the Lung Volume Reduction Coil (LVRC) for the treatment of patients with emphysema in multiple centers.

ELIGIBILITY:
Inclusion Criteria:

* Greater than or equal to 35 years of age
* bilateral heterogenous emphysema
* Patient has stopped smoking for a minimum of 8 weeks
* Read, understood and signed the Informed consent form

Exclusion Criteria:

* Patient has a history of recurrent significant respirator infection
* Patient has an inability to walk > 140 meters
* Patient has evidence of other disease that may compromise survival such as lung cancer, renal failure, etc
* Patient is pregnant or lactating
* Patient has clinical significant bronchiectasis
* Patient has had previous LVR surgery, lung transplant or lobectomy
* Patient has been involved in other pulmonary drug studies within 30 days prior to this study

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2009-12; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
St. George's Respiratory Questionnaire | 6 months
  Symptomatic improvement in St. George's Respiratory Questionnaire (SGRQ) from Baseline

CONTACTS AND LOCATIONS:
Locations (11):
- France (3):
  - CHU de Nice - Hospital Pasteur, Nice
  - Gaetan Deslee, Reims
  - CHRU de Strasbourg-NHC, Strasbourg
- Germany (7):
  - Campus Charite Mitte, Berlin
  - Klinikum Donaustauf, Donaustauf
  - Asklepios, Gauting
  - Thoraxklinik, Heidelberg
  - Lungenklinik, Hemer
  - Krankenhaus von Roten Kreuz, Stuttgart
  - UKT University Hospital, Teubingen
- University Medical Center Groningen, Groningen, Netherlands

REFERENCES:
- [Derived] Hartman JE, Klooster K, Gortzak K, ten Hacken NH, Slebos DJ. Long-term follow-up after bronchoscopic lung volume reduction treatment with coils in patients with severe emphysema. Respirology. 2015 Feb;20(2):319-26. doi: 10.1111/resp.12435. Epub 2014 Nov 23. PMID 25418910
- [Derived] Deslee G, Klooster K, Hetzel M, Stanzel F, Kessler R, Marquette CH, Witt C, Blaas S, Gesierich W, Herth FJ, Hetzel J, van Rikxoort EM, Slebos DJ. Lung volume reduction coil treatment for patients with severe emphysema: a European multicentre trial. Thorax. 2014 Nov;69(11):980-6. doi: 10.1136/thoraxjnl-2014-205221. Epub 2014 Jun 2. PMID 24891327